CLINICAL TRIAL: NCT03089229
Title: A Study to Evaluate the Efficacy and Safety of HAT01H, a Novel Topical Therapeutic: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Efficacy and Safety of HAT01H in Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Haus Bioceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCTP17MD11
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Topical Cream; Novel
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Sponsor will send all washout and test products in compliance with current Good Manufacturing Practices directly to the clinical facility prior to the start of the study. Study procedures will be in place to ensure double-blind administration of study treatments. Access to the randomization code will be strictly controlled. The quantity of all study material shipped to the clinical facility will be documented on the shipping and receiving form included within the shipment. Due to the objectives of the study, the identity of test and control treatments will not be known to investigators, care provider, outcomes assessor, research staff, or patients. Packaging and labeling of test and control treatments will be identical to maintain the blind. Products will be identified with the codes generated by the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HAT01H cream (Experimental): HAT01H medicated cream will come in a blinded tube. This topical medicated cream will be applied once in the morning and once in the evening at least 8 hours apart to all lesions. Treatment will continue daily until next visit.
  Interventions: Drug: HAT01H Cream
- Vehicle cream (Placebo Comparator): Vehicle cream will come in a blinded tube. This topical medicated vehicle will be applied once in the morning and once in the evening at least 8 hours apart to all lesions. Treatment will continue daily until next visit.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: HAT01H Cream — HAT01H Cream will be applied twice daily. The research team will provide instructions for the correct application of the treatment. If a lesion disappears, patients will continue applying the cream twice daily to the area. No additional creams, lotions or soaps other than provided test products will be allowed throughout the duration of the study.
  Other Names: HAT01H
  Arms: HAT01H cream
Drug: Vehicle Cream — Vehicle Cream will be applied twice daily. The research team will provide instructions for the correct application of the treatment. If a lesion disappears, patients will continue applying the cream twice daily to the area. No additional creams, lotions or soaps other than provided test products will be allowed throughout the duration of the study.
  Other Names: Vehicle
  Arms: Vehicle cream

SUMMARY:
Atopic dermatitis (AD) is a chronic inflammatory skin disease characterized by a disturbance of epidermal-barrier function that results in intensely pruritic subacute and chronic eczematous plaques. The current therapy of AD is reactive, where the flares are treated through symptomatic management with topical corticosteroids and calcineurin inhibitors. Given that these medications have long-term side-effects, and given the chronically relapsing immunopathogenic nature of AD, there is an imperative need for safer anti-inflammatory medications. Haus Bioceuticals (Haus) has developed a novel topical treatment for eczema/atopic dermatitis (AD) denoted HAT01H, and have demonstrated that HAT01H is safe and profoundly effective in the treatment of AD, controlling signs and symptoms in 85% of patients with AD. This study is aimed to further test the efficacy and safety of topical HAT01H in patients with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
This study is a 13 week (91 days) randomized, double-blind, in home use study among 30 male and female subjects with moderate to severe active atopic dermatitis (AD). The study will include subjects with ages 12 - 65 years old inclusive. Group assignments will be balanced by age and disease severity of AD. The study will consist of a 1 week washout period and 12 week treatment phase. During the treatment phase, subject will be provided one of the two test products to use twice daily on all lesions and non-lesional areas as instructed. No additional creams, lotions or soaps other than provided test products will be allowed throughout the duration of the study. Measurements, expert visual assessments and self-assessments will be taken as described below. Safety and tolerability will be evaluated by incidence of AE's (defined per CTCAE), exacerbations, application site reactions/infections, and lab evals. There will also be consumption/compliance checks and dermatological evaluations at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe atopic dermatitis as determined by PGA ≥ 3 and SCORAD > 25
* Males and females, age 12 - 65 years old inclusive

Exclusion Criteria:

* Is currently participating or has participated in another interventional clinical study at this or any other facility in the past 3 months.
* Currently or has been diagnosed or treated for cancer in the past 5 years.
* Requires any topical or systemic medications that could affect the course of their atopic dermatitis during the study period (except inhaled steroids and/or stable antihistamines for asthma or allergies).
* Has a known hypersensitivity to any corticosteroid creams.
* Has any active infections or has used antibiotics in the past 7 days.
* Has any physical attributes or skin conditions that might interfere with clear visual assessments (i.e. cuts, sunburn, birth marks, tattoos, extensive scarring, excessive hair growth or acne)
* Has an immunologic or infectious disease (e.g. hepatitis, tuberculosis, HIV or AIDS, lupus, rheumatoid arthritis) which could place the subject at risk or interfere with the accuracy of the study results.
* Has used any immunosuppressant drugs or immunotherapy within the past 30 days or 5 half-lives.
* Is an employee of the sponsor company or clinical testing site.
* Is dependent on oral medication for any skin disease/condition or could not, in the opinion of the Investigator tolerate the restriction of discontinuing the medicine as required in this study.
* Is currently pregnant or lactating or planning to become pregnant in the next 6 months (using double contraception for prevention).
* Any other condition or factor the Investigator or their duly assigned representative believes may affect the ability of the subject to complete the study or the interpretation of the results.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-03-26 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Scoring of Atopic Dermatitis (SCORAD) score | Baseline to week 12
  The primary efficacy is determined by absolute change from baseline to week 12 in inflammatory SCORAD.

SECONDARY OUTCOMES:
Proportion of patients achieving a Physician's Global Assessment (PGA) score of 0 or 1 | Baseline to week 12
  The secondary efficacy measures is determined by absolute change from baseline to week 12 in PGA
Incidence of treatment emergent Adverse Event | Baseline to week 12
  The secondary efficacy measures also include safety and tolerability (incidence of treatment emergent AE's)

CONTACTS AND LOCATIONS:
Overall Officials: Mukta Sachdev, MD, Principal Investigator — Clinical
Locations (1):
- Clinical Research Pvt Ltd, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: Yes